CLINICAL TRIAL: NCT06835257
Title: Evaluation of the Effect of Different Hemodynamic Managements Throughout Autologous Blood Collection Methods on Pulse Contour Analysis Parameters in Coronary Artery Bypass Graft Surgery
Brief Title: Hemodynamic Management in Autologous Blood Collection for CABG Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muhammed E Aydin, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ATATURK-Hemodynamic
Record Dates: First submitted 2023-08-22; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Bypass Grafting; Acute Normovolemic Hemodilution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute normovolemic hemodilution (Active Comparator): Acute normovolemic hemodilution throughout the autologous blood collection
  Interventions: Procedure: Acute normovolemic hemodilutions
- Vasopressor (Active Comparator): Vasopressor infusion throughout the autologous blood collection
  Interventions: Drug: Vasopressor infusion

INTERVENTIONS:
Procedure: Acute normovolemic hemodilutions — Crystalloid infusion throughout the autologous blood collection (3 ml of crystalloid infusion for every 1 ml of blood)
  Arms: Acute normovolemic hemodilution
Drug: Vasopressor infusion — Vasopressor infusion throughout the autologous blood collection (according to mean arterial pressure)
  Arms: Vasopressor

SUMMARY:
In this study, investigated the hemodynamic differences between patients who underwent acute normovolemic hemodilution during the Autologous Blood Collection procedure in coronary artery bypass graft surgery and those who did not, using hemodynamic and cardiac data obtained by MostCare's pressure recording analytical method (PRAM).

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) surgeries are surgeries in which the need for blood transfusion is high. Allogeneic transfusion and transfusion-related complications have led researchers to use different techniques. Autologous blood collection method is one of the alternative methods used to eliminate the need for transfusion. The acute normovolemic hemodilution technique traditionally applied during autologous blood collection causes hemodilution in CABG surgeries and increases the risk of bleeding in patients. In this study, vasopressor infusion technique was used as an alternative technique to avoid hemodilution during autologous blood collection. These two techniques (Acute normovolemic hemodilution - Vasopressor infusion) applied to maintain hemodynamic stabilization during autologous blood collection were compared with the advanced cardiac and hemodynamic data provided by the pressure recording analytical method. The primary aim of the study was to compare cardiac cycle efficiency (CCE), which is a cardiac performance parameter and provides estimates of the energy spent by the cardiovascular system to maintain hemodynamic balance. Secondary objectives are to compare other advanced hemodynamic and postoperative laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Undergoing isolated coronary artery bypass grafting surgery under general anesthesia
* Invasive blood pressure (radial or femoral) and Mostcare monitoring
* Recruitment after booking for surgery with sufficient time to read, understand and question study patient information prior to attending for surgery
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Refuse to consent to the study
* Arterial wave form distortion
* Cardiac arrhythmia
* Inappropriate identification of the dicrotic notch for any reason
* Hemodynamic instability defined as mean arterial blood pressure < 65 mmHg
* Preoperative requirement of inotrope/vasopressor infusion
* Preoperatively receiving vasoactive drugs
* Patients fitted with an intra-aortic balloon pump
* Patients fitted with Extracorporeal Membrane Oxygenation
* Critically ill patients requiring preoperative intensive care unit
* Presence of intraabdominal hypertension
* New York Heart Association Class 3-4 heart failure
* Congestive heart failure with ejection fraction < 35%
* Glomerular filtration rate < 30 ml/min/1.73 m2
* Ongoing renal replacement therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the effects of different techniques used for autologous blood collection on Cardiac Cycle Efficiency (CCE) changes obtained by pulse contour analysis. | From the beginning to the end of autologous blood collection (in the first 30 minutes of surgery)
  Difference of Cardiac Cycle Efficiency(CCE) PRAM parameters between patients

SECONDARY OUTCOMES:
Comparison of the Contractility (dP/dtmax mmHg/msec), Stroke Volume Index (SVI mL/m2), Cardiac Power Index (CPI W/m2), Arterial Elastance (Ea mmHg/mL), Stroke Volume Variation (SVV %), Pulse Pressure Variation (PPV %) changes | From the beginning to the end of autologous blood collection (in the first 30 minutes of surgery)
  Difference of other PRAM and traditional hemodynamic parameters between patients

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ataturk University, Erzurum, Yakutiye
  - Ataturk University, Erzurum

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bennett-Guerrero E, Zhao Y, O'Brien SM, Ferguson TB Jr, Peterson ED, Gammie JS, Song HK. Variation in use of blood transfusion in coronary artery bypass graft surgery. JAMA. 2010 Oct 13;304(14):1568-75. doi: 10.1001/jama.2010.1406. PMID 20940382
- [Background] Coursin DB, Monk TG. Extreme normovolemic hemodilution: how low can you go and other alternatives to transfusion? Crit Care Med. 2001 Apr;29(4):908-10. doi: 10.1097/00003246-200104000-00051. No abstract available. PMID 11373498
- [Background] Romano SM, Pistolesi M. Assessment of cardiac output from systemic arterial pressure in humans. Crit Care Med. 2002 Aug;30(8):1834-41. doi: 10.1097/00003246-200208000-00027. PMID 12163802